CLINICAL TRIAL: NCT00708799
Title: Efficacy of Macrolide Immunomodulation in Severe Sepsis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety evaluation due to recent publications.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Northwestern University Feinberg School of Medicine (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VISN 17-001; 5K23HL096054-03 (NIH); UHS#20151 (Other: UTHSCSA/South Texas Veterans Health Care System)
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Standard antibiotic therapy +Azithromycin 500 mg intravenously daily for 5 days
  Interventions: Other: Azithromycin on admission - not enrolled in the RCT
- Arm 2 (No Intervention): Standard antibiotic therapy

INTERVENTIONS:
Other: Azithromycin on admission - not enrolled in the RCT — One dose of azithromycin prior to inclusion to the RCT
  Other Names: Arm 3
  Arms: Arm 1

SUMMARY:
The purpose of this study is to determine whether macrolide treatment of patients with severe sepsis has an advantageous immunomodulatory and clinical effect compared to severe septic patients without macrolide therapy. Our main hypothesis is macrolide use in addition to standard therapy in severe septic patients has an advantageous immunomodulatory and clinical effect compared to patients with severe sepsis not treated with a macrolide.

DETAILED DESCRIPTION:
In recent studies, the significant effects of macrolide antibiotics (azithromycin) on immune response, unrelated to their anti-microbial properties, have been appreciated. Clinical trials of macrolides added to -lactams in bacteremic Streptococcus pneumoniae community-acquired pneumonia (CAP) have consistently demonstrated an absolute risk reduction in mortality of 15% in most populations. Several cytokines including tumor necrosis factor (TNF) interleukin (IL) -1 and IL-8 which are generally proinflammatory and IL-6 and IL-10, which tend to be anti-inflammatory have been associated with sepsis. TNF is a cytokine that for a number of reasons is thought to play a central role in the pathogenesis of sepsis and septic shock. TNF concentrations are increased during clinical and experimental sepsis and increasing concentrations and especially persistence of high concentrations of TNF during sepsis are associated with decreased survival. Therefore, our primary aim is to determine whether macrolide treatment of patients with severe sepsis has an advantageous immunomodulatory and clinical effect compared to severe septic patients without macrolide therapy. Our main hypothesis is macrolide use in addition to standard therapy in severe septic patients has an advantageous immunomodulatory and clinical effect compared to patients with severe sepsis not treated with a macrolide.

ELIGIBILITY:
Inclusion Criteria:

1. Subject, or legal representative, has given written informed consent.
2. 18 years of age or older.
3. SIRS is defined as two or more of:

   * Temperature > 38o C or < 36oC
   * Heart rate > 90 beats/min
   * Respiratory rate > 20 breaths/min or PaCO2< 32mmHg
   * White blood cell count > 12.000/mm3; < 4000/mm3; or > 10% immature (band) forms.
4. Presence of a suspected or proven infection. Patients with suspected infection must have evidence of an infection, such as white blood cells in a normally sterile body fluid, perforated viscus, chest x-ray consistent with pneumonia and associated with purulent sputum production, or a clinical syndrome associated with a high probability of infection (for example, purpura fulminans or ascending cholangitis).
5. Presence of one or more sepsis-associated organ failure. The onset of the first sepsis-associated organ failure must occur within the 48-hour period immediately preceding initiation of study drug infusion. A patient must have an organ failure attributable to the sepsis episode. The organ failure must be newly developed and not explained by underlying disease processes or by effects of concomitant therapy.

   * Cardiovascular: An arterial systolic blood pressure (SBP) of 90 mm Hg or a mean arterial pressure (MAP) 70 mm Hg for at least 1 hour despite adequate fluid resuscitation, adequate intravascular volume status, or the need for vasopressors to maintain SBP 90 mm Hg or MAP 70 mm Hg.
   * Renal: Average urine output <0.5 mL/kg/h for 1 hour despite adequate fluid resuscitation
   * Respiratory: Evidence of acute pulmonary dysfunction PaO2/FiO2 300 and, clinical exam or pulmonary capillary wedge pressure not suggestive of volume overload. If pneumonia is the suspected site of infection, the patient must have a PaO2/FiO2 200.
   * Hematology: Platelet count <80,000/mm3 or a 50% decrease in platelet count from the highest value recorded over the last 3 days.
   * Unexplained metabolic acidosis: Defined by (1) pH 7.30 or base deficit 5.0 mEq/L or (2) plasma lactate level >1.5 times the upper limit of normal.

Adequate fluid resuscitation or adequate intravascular volume is defined as either pulmonary arterial wedge pressure 12 mm Hg or central venous pressure 8 mm Hg. Vasopressors is defined as dopamine 5 g/kg/min or any dose of norepinephrine, epinephrine, or phenylephrine. Dobutamine is not considered a vasopressor.

Exclusion Criteria:

1. Macrolide therapy indicated for clinical condition. If after randomization, the treating physician determines that a macrolide is indicated and no other alternative antibiotic is appropriate, the patient will be excluded from the trial. However, if only one dose of azithromycin had been given and the treating physician decided to stop it, azithromycin might be administered.
2. Known allergy to macrolides.
3. Prolonged QT syndrome or on medications with increased risk of QT prolongation.
4. Pregnant or lactating.

Immunosuppression as defined by:

1. Chemotherapy within the last 30 days,
2. Leukemia or lymphoma which is not in remission,
3. Solid organ or bone marrow/stem cell transplant,
4. Human Immunodeficiency Virus infection with CD4 count < 200 cells/mm3,
5. Chronic corticosteroid use equivalent to > 10 mg prednisone per day,
6. Patient or family decision to limit ICU care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-11 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in cytokines expression | Between admission and day five of treatment

SECONDARY OUTCOMES:
28-day mortality | 28 days or discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marcos I Restrepo, MD BA MSc, Principal Investigator — South Texas Health Care System, San Antonio, TX
Locations (1):
- South Texas Health Care System, San Antonio, TX, San Antonio, Texas, United States

REFERENCES:
- [Derived] Lopes Junior E, Leite HP, Pinho Franco MDC, Konstantyner T. Association of selenium status with endothelial activation during acute systemic inflammation in children. Clin Nutr ESPEN. 2022 Feb;47:367-374. doi: 10.1016/j.clnesp.2021.11.007. Epub 2021 Nov 14. PMID 35063229